CLINICAL TRIAL: NCT07402369
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Phase II Clinical Study to Explore the Efficacy and Safety of Different Doses of CMS-D002 Capsule in Participants With Uterine Fibroids Associated With Menorrhagia
Brief Title: Phase II Study of CMS-D002 Capsule for Uterine Fibroids With Menorrhagia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Kangzhe Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D002-02-001
Record Dates: First submitted 2026-02-03; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Uterine Fibroids With Menorrhagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CMS-D002 Capsules 10 mg (Experimental): CMS-D002 Capsules 10 mg, QD
  Interventions: Drug: CMS-D002 Capsules 10 mg
- CMS-D002 Capsules 25 mg (Experimental): CMS-D002 Capsules 25 mg, QD
  Interventions: Drug: CMS-D002 Capsules 25 mg
- CMS-D002 Capsules 50 mg (Experimental): CMS-D002 Capsules 50 mg, QD
  Interventions: Drug: CMS-D002 Capsules 50 mg
- Placebo (Placebo Comparator): Placebo, QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CMS-D002 Capsules 10 mg — CMS-D002 Capsules 10 mg, QD
  Arms: CMS-D002 Capsules 10 mg
Drug: CMS-D002 Capsules 25 mg — CMS-D002 Capsules 25 mg, QD
  Arms: CMS-D002 Capsules 25 mg
Drug: CMS-D002 Capsules 50 mg — CMS-D002 Capsules 50 mg, QD
  Arms: CMS-D002 Capsules 50 mg
Drug: Placebo — Placebo, QD
  Arms: Placebo

SUMMARY:
Objective This study evaluates whether CMS-D002 capsules are effective in treating menorrhagia in participants with uterine fibroids associated with menorrhagia. The primary outcome is the percentage of participants who achieve menstrual blood loss <80 mL and a reduction of ≥50% from baseline.

Study Design This is a placebo-controlled trial. Participants will be randomized to receive either CMS-D002 capsules or a matching placebo for 12 weeks.

Participant Responsibilities Take one CMS-D002 capsule or placebo daily for 12 weeks. Complete an electronic patient diary daily throughout the study to record menstrual bleeding and other symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 1.Non-menopausal females aged 18-50 years.
* 2. Body Mass Index (BMI) ≥ 18 kg/m².
* 3. Participant was diagnosed with uterine fibroids by ultrasound at the time of screening, and has one or more fibroids with a diameter of at least 2 cm (longest diameter).
* 4. Participant's menstrual cycle was ≥ 21 days and ≤ 35 days for the three consecutive months prior to screening, and the menstrual period was ≤ 14 days.
* 5. Menorrhagia due to uterine fibroids.
* 6. Agrees to use the contraceptive method specified in the protocol throughout the entire study period (from signing the informed consent form to 6 months after administration of the investigational drug).

Exclusion Criteria:

* 1. Pregnant or breastfeeding female
* 2. History of childbirth within 6 months prior to screening
* 3. Excessive menstrual bleeding due to other causes or unknown reasons
* 4. Suffering from a severe coagulation disorder (e.g., hemophilia or von Willebrand disease)
* 5. Underwent myomectomy, endometrial ablation, uterine artery embolization, or magnetic resonance-guided focused ultrasound (MRgFUS)/high-intensity focused ultrasound (HIFUS) ablation within 6 months prior to screening
* 6. Underwent endometrial ablation within one year prior to screening
* 7. Severe infection, severe trauma, or major surgery within the 6 months prior to screening.
* 8. History of malignant tumors within the 5 years prior to screening (excluding cured skin cancer, basal cell carcinoma, and other localized malignant tumors).
* 9. Current or past (within 1 year) history of alcohol or drug abuse (including analgesic abuse).
* 10. Currently participating in other research projects and having used the investigational drug/treatment within 12 weeks prior to administration.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with menstrual bleeding < 80 mL and a reduction of ≥50% from baseline | 12 weeks

SECONDARY OUTCOMES:
Changes in maximum fibroid volume from baseline | 12weeks
Changes in uterine volume from baseline | 12weeks
Percentage of participants without menstrual bleeding or spotting | 4、8、12 weeks
Changes in hemoglobin concentration from baseline | 4、8、12 weeks
Changes in uterine fibroid symptoms and quality of life questionnaire (UFS-QoL) scores from baseline | 12 weeks
  Transformed score ranges from 0 to 100 based on Likert scale (None of time, a little of time, some of the time, most of the time and all of the time). Lower score indicates minimal symptom severity and higher score indicates maximum symptom severity. A negative change from baseline indicates improvement.
Adverse events | Up to week 18

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
To protect the privacy and confidentiality of study participants, in accordance with ethical guidelines and regulatory requirements, individual participant data (IPD) will not be shared.